CLINICAL TRIAL: NCT06800560
Title: Validating a Novel Instrument Developed by ZOE Ltd. to Measure Menopause-related Symptoms and Quality of Life
Brief Title: The Development, Validation and Application of a Novel Questionnaire Developed by ZOE Ltd Measuring Menopause Symptoms and Subjective Quality of Life
Status: Completed | Type: Observational
Sponsor: Zoe Global Limited (Other)
Responsible Party: Sponsor
Other Study IDs: MenoScale Validation
Record Dates: First submitted 2024-11-12; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Menopause
Keywords: Menopause; Questionnaire Validation; Perimenopause; Postmenopause; Quality of Life; Diet Quality; Menopausal Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- PeriHRT - perimenopausal women currently using hormone replacement therapy: Sub-cohort
  Interventions: Other: MenoScale; Other: Greene Climacteric Scale; Other: RAND 36-Item Health Survey 1.0; Other: PREDICT-FFQ-v1
- Peri - perimenopausal women not using hormone replacement therapy: Sub-cohort
  Interventions: Other: MenoScale; Other: Greene Climacteric Scale; Other: RAND 36-Item Health Survey 1.0; Other: PREDICT-FFQ-v1
- PostHRT - postmenopausal women currently using hormone replacement therapy: Sub-cohort
  Interventions: Other: MenoScale; Other: Greene Climacteric Scale; Other: RAND 36-Item Health Survey 1.0; Other: PREDICT-FFQ-v1
- Post - postmenopausal women not using hormone replacement therapy: Sub-cohort
  Interventions: Other: MenoScale; Other: Greene Climacteric Scale; Other: RAND 36-Item Health Survey 1.0; Other: PREDICT-FFQ-v1

INTERVENTIONS:
Other: MenoScale — Menopause symptom questionnaire
Other: Greene Climacteric Scale — Menopause symptom questionnaire
Other: RAND 36-Item Health Survey 1.0 — Quality of life questionnaire
  Other Names: Short Form 36; SF36; SF-36
Other: PREDICT-FFQ-v1 — Food frequency questionnaire
  Other Names: Food frequency questionnaire; FFQ

SUMMARY:
The MenoScale has been developed from the most common symptoms identified in over 70,000 women to reflect symptom prevalence and user-friendly terminology. It builds and improves on pre-existing scoring tools in four main ways. Firstly, the symptoms assessed are informed by prevalence, as identified from a large cohort. Secondly, the language used to ask about symptoms is modern and accessible as determined through qualitative user research. Thirdly, the impact on quality of life is assessed. Finally, it is already being offered online and completely open access.

The overall aim of this study is to validate the reliability and validity of the MenoScale as an instrument to measure menopausal symptoms and the related subjective impact on quality of life (QoL).

DETAILED DESCRIPTION:
Menopause, a crucial phase in a woman's life, is the disappearance of menstruation for 12 months or longer due to depleted ovarian activity. On average, this stage accounts for over one-third of a woman's lifespan (1). In the United Kingdom (UK), the average age of menopause is 51 years, with the transitional period known as perimenopause occurring from around 45 years (2). As of 2017, there are 13 million menopausal women in the UK, with one third being aged 50 years and over in full time employment (3). It is crucial to have reliable and accessible methods for measuring and tracking symptoms in order to establish medical and lifestyle interventions which may aid in alleviating the burden of these symptoms.

All stages of menopause is accompanied by a wide variety of fluctuating symptoms and subjective experiences of women. Therefore, an online, validated questionnaire offers women the opportunity to monitor their symptoms in real- time which ultimately will: 1) raise awareness by increasing understanding around menopause; 2) empower women to track and manage their menopause themselves; and 3) facilitate conversations by providing data-backed insights to enhance discussions with healthcare providers.

The study has four main objectives:

1. Validate the ability of the MenoScale to measure the prevalence of menopause-related symptoms in comparison to the most widely-used scale in clinical practice.
2. Validate the ability of the MenoScale to measure the impact that symptoms have on overall QoL in comparison to a widely-used QoL scale.
3. Evaluate the test-retest reliability of the MenoScale.
4. Explore relationships between menopause-related symptoms and dietary intake.

RECRUITMENT: Potential participants will be recruited from those who are enrolled onto the ZOE Health Study as well as their friends and family. Potential participants will be contacted via email and provided with a Participant Information Sheet. Participants will be given a minimum of 24 hours after receiving the information sheet to decide whether they would like to take part in the study. Those that would like to take part in the study will be screened using an online form via a secure survey platform and eligible participants will then be asked to provide informed consent.

STUDY DESIGN: Once informed consent has been provided all participants will be asked to complete online versions of a demographics questionnaire (ethnicity, education level, menopause history [age symptoms started, age of last period], HRT usage [type and time period taken]), the MenoScale, Green Climacteric Scale, and the Short Form-36. Participants will also be asked to completed a food frequency questionnaire at baseline only. Participants will be contacted seven days later to repeat the same procedures - except for the demographics, health questionnaire and FFQ. Completion of all questionnaires is expected to take approximately 1 hour at baseline and 15 minutes at follow up.

Biological samples will not be collected in this study, nor will previously collected data be analysed.

The only primary data collection to occur during this study is the following:

* Menopause symptoms questionnaires: MenoScale and Green Climacteric Scale
* Quality of life questionnaire: Short Form 36
* Dietary questionnaire: Predict-Food Frequency Questionnaire-v1
* Demographics questionnaire: ethnicity, BMI, HRT usage, education

References:

1. Bermingham KM, Linenberg I, Hall WL, Kadé K, Franks PW, Davies R, Wolf J, Hadjigeorgiou G, Asnicar F, Segata N, Manson JE, Newson LR, Delahanty LM, Ordovas JM, Chan AT, Spector TD, Valdes AM, Berry SE. Menopause is associated with postprandial metabolism, metabolic health and lifestyle: The ZOE PREDICT study. EBioMedicine. 2022 Nov;85:104303. doi: 10.1016/j.ebiom.2022.104303.
2. Gatenby C, Simpson P. Menopause: Physiology, definitions, and symptoms. Best Pract Res Clin Endocrinol Metab. 2024 Jan;38(1):101855. doi: 10.1016/j.beem.2023.101855.
3. Menopause transition: effects on women's economic participation - GOV.UK [https://www.gov.uk/government/publications/menopause-transition-effects-on-womens-economic-participation]

ELIGIBILITY:
Inclusion Criteria:

Female (sex assigned at birth) Aged 37 - 70 years Peri- or postmenopausal (self-reported)

Exclusion Criteria:

Currently pregnant and/or lactating History of hysterectomy or oophorectomy History of treatment-induced menopause Body mass index of < 18.5 Subject is taking > 5 prescribed medications Subject is unable to provide informed consent online Subject is unable understand the participant information sheet Subject is unable to complete the questionnaires online

Ages: 37 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants for this study will be recruited from the ZOE Health Study, which is a community science app in which participants are actively involved in logging lifestyle and health data, and those who have consented to receiving the ZOE newsletter.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
MenoScale validity for menopause symptoms | Baseline
  The ability of the MenoScale to measure the prevalence of menopause-related symptoms in comparison to the most widely-used scale in clinical practice.

SECONDARY OUTCOMES:
MenoScale validity for quality of life | Baseline
  - The ability of the MenoScale to measure the impact that symptoms have on overall quality of life in comparison to a widely-used quality of life scale.
MenoScale reliability | Baseline and 1 week later
  The reliability of the MenoScale to be repeated and how this compares to the Green Climacteric Scale
Diet quality | Baseline
  Associations between healthy dietary patterns, food groups and menopausal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Berry, PhD, Principal Investigator — King's College London
Locations (1):
- ZOE Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gatenby C, Simpson P. Menopause: Physiology, definitions, and symptoms. Best Pract Res Clin Endocrinol Metab. 2024 Jan;38(1):101855. doi: 10.1016/j.beem.2023.101855. Epub 2023 Dec 21. PMID 38171939
- [Background] Bermingham KM, Linenberg I, Hall WL, Kade K, Franks PW, Davies R, Wolf J, Hadjigeorgiou G, Asnicar F, Segata N, Manson JE, Newson LR, Delahanty LM, Ordovas JM, Chan AT, Spector TD, Valdes AM, Berry SE. Menopause is associated with postprandial metabolism, metabolic health and lifestyle: The ZOE PREDICT study. EBioMedicine. 2022 Nov;85:104303. doi: 10.1016/j.ebiom.2022.104303. Epub 2022 Oct 18. PMID 36270905
- See also: Menopause transition: effects on women's economic participation — https://www.gov.uk/government/publications/menopause-transition-effects-on-womens-economic-participation